CLINICAL TRIAL: NCT02161380
Title: An Open-label Dose Escalation Study of an Adeno-associated Virus Vector (scAAV2-P1ND4v2) for Gene Therapy of Leber's Hereditary Optic Neuropathy (LHON) Caused by the G11778A Mutation in Mitochondrial DNA
Brief Title: Safety Study of an Adeno-associated Virus Vector for Gene Therapy of Leber's Hereditary Optic Neuropathy
Acronym: LHON
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Byron Lam (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor-Investigator, Byron Lam, Greene Professor of Ophthalmology, University of Miami
Organization: University of Miami (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20140248; 1U10EY023558-01A1 (NIH)
Record Dates: First submitted 2014-06-06; First posted 2014-06-11 (Estimated); Results first posted 2024-08-07 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Leber's Hereditary Optic Neuropathy
Keywords: Gene therapy; Mitochondrial Genes; Leber's; AAV2 Viral vectors
MeSH Terms: conditions — Optic Atrophy, Hereditary, Leber | interventions — Matrilin Proteins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Low-dose (1.18x10e9 vg) (Experimental): Participants with Chronic Bilateral Severe Vision Loss were administered 200 µL of scAAV2-P1ND4v2 containing a dose of 1.18x10e9 vg.
  Participants with Acute Bilateral Severe Vision Loss were administered 200 µL of scAAV2-P1ND4v2 containing a dose of 1.18x10e9 vg.
  Participants with Acute Unilateral Severe Vision Loss were administered 200 µL of scAAV2-P1ND4v2 containing a dose of 1.18x10e9 vg
  Interventions: Drug: injection of scAAV2-P1ND4v2 1.18x10e9 vg (Low),
- Medium dose (5.81x10e9 vg) (Experimental): Participants with Chronic Bilateral Severe Vision Loss were administered 200 µL of scAAV2-P1ND4v2 containing a dose of 5.81x10e9 vg.
  Participants with Acute Bilateral Severe Vision Loss were administered 200 µL of scAAV2-P1ND4v2 containing a dose of 5.81x10e9 vg.
  Participants with Acute Unilateral Severe Vision Loss were administered 200 µL of scAAV2-P1ND4v2 containing a dose of 5.81x10e9 vg.
  Interventions: Drug: injection of scAAV2-P1ND4v2 5.81 X10e9 vg (Med)
- High dose (2.40x10e10 vg) (Experimental): Participants with Chronic Bilateral Severe Vision Loss were administered 100 µL of scAAV2-P1ND4v2 containing a dose of 2.40x10e10 vg.
  Interventions: Drug: injection of scAAV2-P1ND4v2 2.4 X10e10vg (High)
- Higher dose (1x10e11vg) (Experimental): Participants with Chronic Bilateral Severe Vision Loss were administered 100 µL of scAAV2-P1ND4v2 containing a dose of 1x10e11vg.
  Participants with Acute Bilateral Severe Vision Loss were administered 100 µL of scAAV2-P1ND4v2 containing a dose of 1x10e11vg.
  Participants with Acute Unilateral Severe Vision Loss were administered 100 µL of scAAV2-P1ND4v2 containing a dose of 1x10e11vg.
  Interventions: Drug: injection of scAAV2-P1ND4v2 1.0 X10e11vg (Higher)

INTERVENTIONS:
Drug: injection of scAAV2-P1ND4v2 1.18x10e9 vg (Low), — injection of Total Volume of each intravitreal injection is 200 µL
  Other Names: AAV-ND4
  Arms: Low-dose (1.18x10e9 vg)
Drug: injection of scAAV2-P1ND4v2 5.81 X10e9 vg (Med) — injection of Total Volume of each intravitreal injection is 200 µL
  Other Names: AAV-ND4
  Arms: Medium dose (5.81x10e9 vg)
Drug: injection of scAAV2-P1ND4v2 2.4 X10e10vg (High) — injection of Total Volume of each intravitreal injection is 100 µL
  Other Names: AAV-ND4
  Arms: High dose (2.40x10e10 vg)
Drug: injection of scAAV2-P1ND4v2 1.0 X10e11vg (Higher) — injection of Total Volume of each intravitreal injection is 100 µL
  Other Names: AAV-ND4
  Arms: Higher dose (1x10e11vg)

SUMMARY:
The study is a dose-escalation study, phase 1. The objective of this proposed clinical trial is to evaluate the safety of mitochondrially targeted ND4 gene therapy with the adeno-associated viral vector in appropriate LHON patients.

DETAILED DESCRIPTION:
The purpose of this dose-escalation study is to assess the safety and tolerability of scAAV2-P1ND4v2 (abbreviated as AAV-ND4) gene replacement therapy in subjects confirmed with the G11778A mutation in mtDNA responsible for Leber's Hereditary Optic Neuropathy. Ocular and systemic toxicity will be assessed following vector administration to determine if there are adverse changes that may be associated with vector administration.

This first-in-man (FIM) clinical trial will assess the safety, tolerability, and potential efficacy of a single intravitreal injection in patient groups reflecting the acute, pre-symptomatic, and chronic stages and manifestation of the LHON disease.

ELIGIBILITY:
Inclusion Criteria:

1. Age 15 or older;
2. Patients with LHON and the G11778A mitochondrial DNA mutation. A previous CLIA-certified genetic lab result showing the LHON G11778A mutation will be accepted for inclusion;
3. Ability to perform tests of visual and retinal function;
4. Ability to comply with research procedures;
5. Able and willing to provide informed consent before undergoing any study-related procedures.
6. Good general health as based on the investigator's assessment of the history, physical examination, and laboratory testing performed at the baseline examination.

Exclusion Criteria:

1. Unwilling or unable to give consent,
2. Unable or unlikely to return for scheduled protocol visits
3. Pregnant or nursing women or unwillingness for subject with childbearing potential to use contraception during the first year of the study.
4. Optic disc drusen on exam or in previous history.
5. Ocular diseases or visual dysfunction conditions other than refractive error (e.g. amblyopia, glaucoma, etc.) in the eye selected for the injection.
6. Previous eye surgery in the eye selected for injection.
7. Aspartate transaminase (AST)/alanine transaminase (ALT) >5.0 x upper limit of normal (ULN); Total bilirubin >3 x ULN; Hemoglobin < 8 g/dL; neutrophil count <1.0 x 109/L; or platelet count < 50 x 109/L

   a) Any laboratory screening test that meets the abnormality criteria stated above can be repeated once between Baseline one to Baseline 2.
8. Type I diabetes or the presence of diabetic retinopathy
9. History of neurodegenerative conditions (e.g. multiple sclerosis, neuromyelitis optica, Parkinson's disease)
10. History of autoimmune conditions (e.g. systemic lupus erythematosus)
11. Systemic diseases having ocular manifestations likely to confound assessment of study results. History of cancer within five years other than localized basal or squamous cell carcinoma not near the orbital area. Patients with a prior history of cancer will need documentation from their cancer specialist that the cancer was cured at least 5 years before study entry.
12. Allergy to pupil dilating drops or narrow angles precluding safe dilation.
13. No Light Perception (NLP) vision in either eye.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-07-14 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2025-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Byron Lam, MD, Principal Investigator — Bascom Palmer Eye Institute, Miller School of Medicine, University of Miami, Miami, FL 33136
Locations (1):
- Bascom Palmer Eye Institute, University of Miami, Miami, Florida, United States

REFERENCES:
- [Result] Feuer WJ, Schiffman JC, Davis JL, Porciatti V, Gonzalez P, Koilkonda RD, Yuan H, Lalwani A, Lam BL, Guy J. Gene Therapy for Leber Hereditary Optic Neuropathy: Initial Results. Ophthalmology. 2016 Mar;123(3):558-70. doi: 10.1016/j.ophtha.2015.10.025. Epub 2015 Nov 19. PMID 26606867
- [Result] Guy J, Feuer WJ, Davis JL, Porciatti V, Gonzalez PJ, Koilkonda RD, Yuan H, Hauswirth WW, Lam BL. Gene Therapy for Leber Hereditary Optic Neuropathy: Low- and Medium-Dose Visual Results. Ophthalmology. 2017 Nov;124(11):1621-1634. doi: 10.1016/j.ophtha.2017.05.016. Epub 2017 Jun 21. PMID 28647203
- [Result] Lam BL, Feuer WJ, Davis JL, Porciatti V, Yu H, Levy RB, Vanner E, Guy J. Leber Hereditary Optic Neuropathy Gene Therapy: Adverse Events and Visual Acuity Results of All Patient Groups. Am J Ophthalmol. 2022 Sep;241:262-271. doi: 10.1016/j.ajo.2022.02.023. Epub 2022 Mar 7. PMID 35271811
- [Result] Lam BL, Feuer WJ, Porciatti V, Davis JL, Zheng DD, Vanner EA, Savatovsky EJ, Alba DE, Guy J. Leber Hereditary Optic Neuropathy Gene Therapy: Longitudinal Relationships Among Visual Function and Anatomical Measures. Am J Ophthalmol. 2024 Jan;257:113-128. doi: 10.1016/j.ajo.2023.09.005. Epub 2023 Sep 15. PMID 37716450
- [Result] Porciatti V, Alba DE, Feuer WJ, Davis J, Guy J, Lam BL. The Relationship Between Stage of Leber's Hereditary Optic Neuropathy and Pattern Electroretinogram Latency. Transl Vis Sci Technol. 2022 Mar 2;11(3):31. doi: 10.1167/tvst.11.3.31. PMID 35344016
- [Result] Lam BL. Leber hereditary optic neuropathy gene therapy. Curr Opin Ophthalmol. 2024 May 1;35(3):244-251. doi: 10.1097/ICU.0000000000001028. Epub 2023 Dec 20. PMID 38117686
- [Result] Lam BL, Burke SP, Wang MX, Nadayil GA, Rosa PR, Gregori G, Feuer WJ, Cuprill-Nilson S, Vandenbroucke R, Zhang X, Guy J. Macular Retinal Sublayer Thicknesses in G11778A Leber Hereditary Optic Neuropathy. Ophthalmic Surg Lasers Imaging Retina. 2016 Sep 1;47(9):802-10. doi: 10.3928/23258160-20160901-02. PMID 27631475
- [Result] Koilkonda R, Yu H, Talla V, Porciatti V, Feuer WJ, Hauswirth WW, Chiodo V, Erger KE, Boye SL, Lewin AS, Conlon TJ, Renner L, Neuringer M, Detrisac C, Guy J. LHON gene therapy vector prevents visual loss and optic neuropathy induced by G11778A mutant mitochondrial DNA: biodistribution and toxicology profile. Invest Ophthalmol Vis Sci. 2014 Oct 23;55(12):7739-53. doi: 10.1167/iovs.14-15388. PMID 25342621
- [Result] Guy J, Feuer WJ, Porciatti V, Schiffman J, Abukhalil F, Vandenbroucke R, Rosa PR, Lam BL. Retinal ganglion cell dysfunction in asymptomatic G11778A: Leber hereditary optic neuropathy. Invest Ophthalmol Vis Sci. 2014 Feb 10;55(2):841-8. doi: 10.1167/iovs.13-13365. PMID 24398093
- [Result] Koilkonda RD, Yu H, Chou TH, Feuer WJ, Ruggeri M, Porciatti V, Tse D, Hauswirth WW, Chiodo V, Boye SL, Lewin AS, Neuringer M, Renner L, Guy J. Safety and effects of the vector for the Leber hereditary optic neuropathy gene therapy clinical trial. JAMA Ophthalmol. 2014 Apr 1;132(4):409-20. doi: 10.1001/jamaophthalmol.2013.7630. PMID 24457989
- [Derived] Davis JL. The Blunt End: Surgical Challenges of Gene Therapy for Inherited Retinal Diseases. Am J Ophthalmol. 2018 Dec;196:xxv-xxix. doi: 10.1016/j.ajo.2018.08.038. Epub 2018 Sep 5. PMID 30194931
- See also: Bascom Palmer News — http://bascompalmer.org/news

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at Bascom Palmer Eye Institute (Single institution study) in Florida, United States(US) from 14 July 2014 to 18 Nov 2020.
Pre-assignment Details: A total of 28 participants with G11778A Leber Hereditary Optic Neuropathy (LHON) were enrolled in the study. They were distributed in the following groups: chronic bilateral visual loss > 12 months (group 1, n=11), acute bilateral visual loss < 12 months (group 2, n=9), or unilateral visual loss (group 3, n=8). Each participant received a unilateral intravitreal injection. Group 1 was treated with low, medium, high and higher dose, group 2 and 3 were treated with low, medium, or higher dose.
Groups:
- Low-dose (1.18x10e9 vg): Participants with Chronic Bilateral Severe Vision Loss were administered 200 µL of scAAV2-P1ND4v2 containing a dose of 1.18x10e9 vg.
  Participants with Acute Bilateral Severe Vision Loss were administered 200 µL of scAAV2-P1ND4v2 containing a dose of 1.18x10e9 vg.
  Participants with Acute Unilateral Severe Vision Loss were administered were administrated 200 µL of scAAV2-P1ND4v2 containing a dose of 1.18x10e9 vg.
- Medium Dose (5.81x10e9 vg): Participants with Chronic Bilateral Severe Vision Loss were administered 200 µL of scAAV2-P1ND4v2 containing a dose of 5.81x10e9 vg.
  Participants with Acute Bilateral Severe Vision Loss were administered 200 µL of scAAV2-P1ND4v2 containing a dose of 5.81x10e9 vg.
  Participants with Acute Unilateral Severe Vision Loss were administered were administrated 200 µL of scAAV2-P1ND4v2 containing a dose of 5.81x10e9 vg.
- Higher Dose (1x10e11vg): Participants with Chronic Bilateral Severe Vision Loss were administered 100 µL of scAAV2-P1ND4v2 containing a dose of 1x10e11vg.
  Participants with Acute Bilateral Severe Vision Loss were administrated 100 µL of scAAV2-P1ND4v2 containing a dose of 1x10e11vg.
  Participants with Acute Unilateral Severe Vision Loss were administered 100 µL of scAAV2-P1ND4v2 containing a dose of 1x10e11vg.
Period: Overall Study
Arm/Group | Low-dose (1.18x10e9 vg) | Medium Dose (5.81x10e9 vg) | High Dose (2.40x10e10 vg) | Higher Dose (1x10e11vg)
Started | 9 | 9 | 3 | 7
Chronic Bilateral | 3 | 3 | 3 | 2
Acute Bilateral | 3 | 3 | 0 | 3
Acute Unilateral | 3 | 3 | 0 | 2
Completed | 9 | 8 | 3 | 7
Not Completed | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Medium Dose (5.81x10e9 vg): Participants with Chronic Bilateral Severe Vision Loss were administered 200 µL of scAAV2-P1ND4v2 containing a dose of 5.81x10e9 vg.
  Participants with Acute Bilateral Severe Vision Loss were administrated 200 µL of scAAV2-P1ND4v2 containing a dose of 5.81x10e9 vg.
  Participants with Acute Unilateral Severe Vision Loss were administered 200 µL of scAAV2-P1ND4v2 containing a dose of 5.81x10e9 vg.
- Total: Total of all reporting groups
Arm/Group | Low-dose (1.18x10e9 vg) | Medium Dose (5.81x10e9 vg) | High Dose (2.40x10e10 vg) | Higher Dose (1x10e11vg) | Total
Number analyzed (Participants) | 9 | 9 | 3 | 7 | 28
Age, Continuous [Mean (Full Range); unit: years] | 36.44 [19 to 56] | 25.22 [16 to 33] | 25.66 [19 to 33] | 34.14 [16 to 51] | 31.1 [16 to 56]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 0 | 1 | 5
  Male | 8 | 6 | 3 | 6 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 2 | 4
  Not Hispanic or Latino | 8 | 9 | 2 | 5 | 24
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 9 | 8 | 3 | 7 | 27
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Treatment Related Adverse Events
Description: Number of treatment-related adverse events will be assessed as per investigator with respective to relationship to the investigative product.
Time Frame: 3 years
Population: One subject for medium dose was a loss to follow up after month 06. One subject for low dose missed visits for month 12, month 24 and month 36
Measure: Count of Participants; unit: Participants
Arm/Group | Low-dose (1.18x10e9 vg) | Medium Dose (5.81x10e9 vg) | High Dose (2.40x10e10 vg) | Higher Dose (1x10e11vg)
Number analyzed (Participants) | 8 | 8 | 3 | 7
Participants | 1 | 1 | 1 | 5

2. Secondary Outcome: Best-corrected Visual Acuity
Description: Best-corrected visual acuity(BCVA) was tested using the ETDRS Chart. The LogMAR visual acuity scale was adapted from the ETDRS chart to facilitate statistical analysis.
  Longitudinal analyses of BCVA changes at months 12, 24, and 36 versus baseline 2 were performed.
Time Frame: up to 36 months after treatment
Population: One subject for low dose missed visits 12, 24, and 36 months but he completed the majority of the other study visits.
  One subject for medium dose was a loss to follow up after visit 6 months. One subject for higher dose missed a visit 12 months to the COVID-19 pandemic.
Measure: Mean (Standard Deviation); unit: logMar
Arm/Group | Low-dose (1.18x10e9 vg) | Medium Dose (5.81x10e9 vg) | High Dose (2.40x10e10 vg) | Higher Dose (1x10e11vg)
Number analyzed (Participants) | 8 | 8 | 3 | 7
logMar
  12 Months/Chronic Bilateral Severe Vision: number analyzed (Participants) | 3 | 3 | 3 | 2
  12 Months/Chronic Bilateral Severe Vision | 0.03 (0.06) | -0.26 (0.42) | -0.39 (0.25) | -0.007 (0.13)
  12 Months/Acute Bilateral Severe Vision: number analyzed (Participants) | 3 | 2 | 0 | 2
  12 Months/Acute Bilateral Severe Vision | -0.54 (0.43) | 0.07 (0.18) |  | 0.26 (0.23)
  12 Months/Acute Unilateral Severe Vision: number analyzed (Participants) | 2 | 3 | 0 | 2
  12 Months/Acute Unilateral Severe Vision | 1.08 (0.17) | 1.29 (0.53) |  | 1.09 (0.30)
  24 Months/Chronic Bilateral Severe Vision: number analyzed (Participants) | 3 | 3 | 3 | 2
  24 Months/Chronic Bilateral Severe Vision | -0.19 (0.39) | -0.23 (0.14) | -0.41 (0.23) | -0.07 (0.13)
  24 Months/Acute Bilateral Severe Vision: number analyzed (Participants) | 3 | 2 | 0 | 3
  24 Months/Acute Bilateral Severe Vision | -0.95 (0.61) | -0.23 (0.36) |  | -0.11 (0.46)
  24 Months/Acute Unilateral Severe Vision: number analyzed (Participants) | 2 | 3 | 0 | 2
  24 Months/Acute Unilateral Severe Vision | 0.95 (0.21) | 1.47 (0.44) |  | 0.83 (0.24)
  36 Months/Chronic Bilateral Severe Vision: number analyzed (Participants) | 3 | 3 | 3 | 2
  36 Months/Chronic Bilateral Severe Vision | -0.19 (0.39) | -0.25 (0.39) | -0.40 (0.22) | -0.06 (0.11)
  36 Months/Acute Bilateral Severe Vision: number analyzed (Participants) | 3 | 2 | 0 | 3
  36 Months/Acute Bilateral Severe Vision | -1.01 (0.63) | 0.00 (0.14) |  | -0.16 (0.65)
  36 Months/Acute Unilateral Severe Vision: number analyzed (Participants) | 2 | 3 | 0 | 2
  36 Months/Acute Unilateral Severe Vision | 1.03 (0.24) | 1.49 (0.40) |  | 0.49 (0.24)

ADVERSE EVENTS:
Time Frame: 3 Years
Description: Participants were followed for AE for 3 years. In addition to the SAE definition for clinicaltrial.gov, this study also considered an SAE a decrease in acuity in the injected eye to 0.3 logMAR units (15-letter equivalent) worse than the worst acuity measured in the uninjected fellow eye at the current or any prior study visit.
Arm/Group | Low-dose (1.18x10e9 vg) | Medium Dose (5.81x10e9 vg) | High Dose (2.40x10e10 vg) | Higher Dose (1x10e11vg)
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9 | 0/3 | 0/7
Serious Adverse Events (participants affected / at risk) | 1/9 | 1/9 | 0/3 | 0/7
Other Adverse Events (participants affected / at risk) | 3/9 | 3/9 | 1/3 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low-dose (1.18x10e9 vg) (N=9) | Medium Dose (5.81x10e9 vg) (N=9) | High Dose (2.40x10e10 vg) (N=3) | Higher Dose (1x10e11vg) (N=7)
Visual Acuity Loss (Eye disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) — SAE will be considered a decrease in acuity in the injected eye to 0.3 logMAR units (15-letter equivalent) worse than the worst acuity measured in the uninjected fellow eye at the current or any prior study visit.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low-dose (1.18x10e9 vg) (N=9) | Medium Dose (5.81x10e9 vg) (N=9) | High Dose (2.40x10e10 vg) (N=3) | Higher Dose (1x10e11vg) (N=7)
Uveitis (Eye disorders) | 1 (2) | 1 (1) | 1 (1) | 5 (5) — One participant of Low Dose had two different episodes of Uveitis
Corneal Abrasion (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) — Causality: not related to research. One participant of Higher dose had 2 different adverse events: Corneal abrasion and Uveitis.
Elevated Liver Enzymes (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) — causality: not related to research

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-02-09): https://cdn.clinicaltrials.gov/large-docs/80/NCT02161380/Prot_SAP_000.pdf
  • Informed Consent Form (2020-09-20): https://cdn.clinicaltrials.gov/large-docs/80/NCT02161380/ICF_001.pdf